CLINICAL TRIAL: NCT00384306
Title: Investigation of the Side Effects of Orally Administered Glucocorticoids. An Open Label Study to Investigate the Effects of Orally Administered Prednisolone on Bone Metabolism in Patients With COPD.
Brief Title: Effects Of Oral Prednisolone On Bone Metabolism In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Cambridge (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RES11086
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; prednisolone; bone biopsy; tetracycline labelling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prednisolone

INTERVENTIONS:
Drug: prednisolone

SUMMARY:
The aim of this study is to establish associations between blood and urine markers of bone metabolism with histomorphometric changes (changes in the actual bone structure) resulting from short term oral prednisolone treatment in patients with COPD (chronic obstructive pulmonary disease).

ELIGIBILITY:
Inclusion criteria:

* Females subjects must be unable to have children.
* BMI 19 - 29.9
* Non-smokers, ex-smokers or current light smokers (<10 cigarettes/day)

Exclusion criteria:

* High blood pressure
* Other significant disease
* Use of certain medications (to be decided by the investigator)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Mineral apposition rate Mineralising surface Eroded surface Bone formation rate Osteocalcin levels Serum and urinary deoxypyridinoline | All measured with and without 3 weeks dosing with oral prednisolone

SECONDARY OUTCOMES:
Pharmacokinetic measurements Bone structure and micro computer tomography of bone biopsies Biochemical markers of bone formation, bone break down and hormones | All measured with and without 3 weeks dosing with oral prednisolone

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Centre, Cambridge, United Kingdom